CLINICAL TRIAL: NCT01273610
Title: Tolerability of the Combination of Lapatinib and Trastuzumab in Adults Age 60 or Older With HER2 Positive Locally Advanced or Metastatic Breast Cancer
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: City of Hope Medical Center (Other)
Collaborators: GlaxoSmithKline (Industry); Novartis (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 10112; NCI-2011-00116 (Registry Identifier: NCI CTRP)
Record Dates: First submitted 2011-01-06; First posted 2011-01-10 (Estimated); Results first posted 2022-07-28 (Actual); Last update posted 2025-06-10 (Actual); Status verified 2025-05

CONDITIONS: Breast Neoplasms; HER2/Neu Positive; Geriatric Health Services
Keywords: Breast Neoplasms; HER2 protein, human; Geriatric Health Services; Antineoplastic Agents, Combined; Geriatric Assessment; Pharmacokinetics; Toxicity; Patient Adherence
MeSH Terms: conditions — Breast Neoplasms; Patient Compliance | interventions — Lapatinib; N-(3-chloro-4-((3-fluorobenzyl)oxy)phenyl-6-(5-((methylsulfonyl)ethyl)aminomethyl)-2-furyl)-4-quinazolinamine; Trastuzumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Lapatinib and trastuzumab (Experimental): Patients receive lapatinib ditosylate PO QD and trastuzumab IV once weekly OR once every 3 weeks. Courses repeat every 21 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Lapatinib; Drug: Trastuzumab; Other: laboratory biomarker analysis; Other: pharmacological study

INTERVENTIONS:
Drug: Lapatinib — 250 mg tablets
  Other Names: Tykerb; Tyverb; GSK572016; GW-572016; GW2016
Drug: Trastuzumab — Intravenous injection
  Other Names: Herceptin
Other: laboratory biomarker analysis
  Other Names: Correlative studies
Other: pharmacological study
  Other Names: Correlative studies

SUMMARY:
This phase II trial studies the side effects and how well lapatinib ditosylate and trastuzumab work in treating older patients with human epidermal growth factor receptor 2 (HER2)-positive breast cancer that has spread from where it started to nearby tissue or lymph nodes (locally advanced) or to other parts of the body (metastatic). Lapatinib ditosylate may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth. Monoclonal antibodies, such as trastuzumab, can block tumor growth in different ways. Some block the ability of tumor to grow and spread. Others find tumor cells and help kill them or tumor cancer-killing substances to them. Giving lapatinib ditosylate together with trastuzumab may kill more tumor cells.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES: I. To estimate the safety and tolerability of the combination of trastuzumab and lapatinib (lapatinib ditosylate) in adults age 60 or older with locally advanced or metastatic breast cancer. SECONDARY OBJECTIVES: I. To describe the full toxicity profile including all grades; to estimate the rate of all grades of cardiac toxicity; to estimate the rate of all grades of diarrhea, nausea, and vomiting. II. To describe the pharmacokinetic parameters of lapatinib in older adults. III. To estimate objective response rate and clinical benefit rate as defined by modified Response Evaluation Criteria In Solid Tumors (RECIST) criteria. IV. To estimate median progression-free and overall survival. V. To explore factors other than chronological age that can affect toxicity rates as identified using a cancer-specific geriatric assessment. VI. To estimate rates of adherence to lapatinib in older adults.

OUTLINE: Patients receive lapatinib ditosylate orally (PO) once daily (QD) and trastuzumab intravenously (IV) over 30-90 minutes once weekly OR once every 3 weeks. Courses repeat every 21 days in the absence of disease progression or unacceptable toxicity. After completion of study treatment, patients are followed up for 30 days and then periodically thereafter.

ELIGIBILITY:
Inclusion Criteria:

* Locally advanced or metastatic Her2/Neu positive breast cancer (defined as immunohistochemistry [IHC] 3+ or a fluorescence in situ hybridization [FISH] ratio of >= 2.0); this may be on either a primary tumor or a metastatic site, and there is no time limit from the time the specimen was obtained; locally advanced breast cancer (LABC) includes breast cancers with advanced primary tumors, i.e., large diameter (at least 5 cm) or those with skin and/or chest wall involvement, and advanced regional lymph node involvement; it also includes a rare subgroup, inflammatory breast cancer; in the 2010 American Joint Committee on Cancer and the International Union for Cancer Control (AJCC-UICC) TNM breast cancer staging system, locally advanced breast cancer (LABC) includes patients with stage III disease; this comprises:

  * Advanced primary tumors (tumors > 5 cm in greatest dimension [T3]; direct extension to the chest wall and/or to the skin [T4]: ulceration, skin nodules, and/or edema (including peau d'orange) confined to the same breast, inflammatory breast cancer [IBC, T4d])
  * Advanced regional lymph nodes (ipsilateral level I, II axillary lymph nodes that are clinically fixed or matted or clinically detected internal mammary lymph nodes in the absence of axillary lymph node metastases [N2], ipsilateral infraclavicular [level III axillary] lymph nodes, ipsilateral internal mammary lymph node[s] with axillary lymph nodes, or ipsilateral supraclavicular lymph nodes [N3])
* Both measurable and non-measurable disease are allowed
* Life expectancy of greater than 12 weeks
* Women of child-bearing potential and sexually active men must agree to use adequate contraception prior to study entry for six months following duration of study participation
* Eastern Cooperative Oncology Group (ECOG) performance status =< 2 (Karnofsky performance status >= 60%)
* Hemoglobin >= 10 g/dL (after transfusion if necessary)
* Absolute neutrophil count >= 1,500/mcL
* Platelets >= 100,000/mcL
* Total bilirubin within normal institutional limits
* Aspartate aminotransferase (AST) (serum glutamic oxaloacetic transaminase [SGOT])/aspartate aminotransferase (ALT) (serum glutamate pyruvate transaminase [SGPT]) =< 2.5 X institutional upper limit of normal
* Creatinine clearance >= 30 mL/min as measured using either the Cockcroft-Gault method or 24-hour creatinine clearance
* The above tests must be obtained within 14 days of study treatment
* Cardiac ejection fraction >= 50% as measured by echocardiogram or multiple gated acquisition scan (MUGA) scan
* The ability to swallow and retain oral medication
* Prior treatment with lapatinib or trastuzumab are allowed, provided that the agents have never been given in combination
* Any number of prior cancer treatments, including investigational agents, chemotherapy, hormone therapy, or targeted therapy are allowed
* All patients must have the ability to understand and the willingness to sign a written informed consent

Exclusion Criteria:

* Concurrent investigational treatment, chemotherapy, or targeted therapy; prior chemotherapy, hormonal therapy, targeted therapy, and investigational agents are allowed but all toxicities grade >= 2 must have resolved by the time of study commencement (except alopecia)
* Unstable or symptomatic brain metastases (however, patients with stable or treated brain metastases who do not require steroids at doses above those permitted for control of symptoms may be enrolled)
* History of allergic reactions attributed to compounds of similar chemical or biological composition to lapatinib or trastuzumab; however, patients with a history of infusion reaction to trastuzumab which was controlled with premedication on subsequent infusions without a recurring infusion reaction are eligible
* Concomitant medications listed are prohibited; inhibitors or inducers of cytochrome P450 3A4 (CYP3A4) not listed can be used with caution
* Ongoing or active infection (including human immunodeficiency virus [HIV]) or psychiatric illness/social situations that would limit compliance with study requirements
* Inability to take oral medication
* Malabsorption syndrome, (prior surgical procedures affecting absorption), or inflammatory gastrointestinal (GI) disease (e.g., Crohn's, ulcerative colitis) which in the opinion of the study coordinator is likely to limit normal absorption of the drug
* Current active hepatic or biliary disease (with the exception of patients with Gilbert's syndrome, asymptomatic gallstones, liver metastases, or stable chronic liver disease per investigator assessment)
* Active cardiac disease, defined as (but not limited to):

  * History of documented congestive heart failure (CHF) or systolic dysfunction (left ventricular ejection fraction [LVEF] < 50%)
  * High-risk uncontrolled arrhythmias (ventricular tachycardia, high-grade atrio-ventricular [AV]-block, supraventricular tachycardias which are not adequately rate-controlled)
  * Angina pectoris requiring antianginal medications
  * Evidence of transmural infarction on electrocardiogram (ECG)
  * Clinically significant valvular heart disease
  * Poorly controlled hypertension (e.g. systolic > 180 mm HG or diastolic > 100 mm Hg)
  * Any other cardiac condition, which in the opinion of the treating physician would make this protocol unreasonably hazardous for the patient
* Subjects who, in the opinion of the investigator, may not be able to comply with the safety monitoring requirements of the study are not eligible

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2011-04-20 (Actual); Primary Completion 2018-02-22 (Actual); Study Completion 2026-05-19 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Daneng Li, MD, Principal Investigator — City of Hope Medical Center
Locations (8):
- United States (8):
  - City of Hope Medical Center, Duarte, California
  - City of Hope Antelope Valley, Lancaster, California
  - South Pasadena Cancer Center, Pasadena, California
  - Roswell Park Cancer Institute, Buffalo, New York
  - Lineberger Comprehensive Cancer Center, University of North Carolina, Chapel Hill, North Carolina
  - Duke University Medical Center, Durham, North Carolina
  - Case Western Reserve University, Cleveland, Ohio
  - Thomas Jefferson University, Philadelphia, Pennsylvania

REFERENCES:
- [Background] Hurria A, Gupta S, Zauderer M, Zuckerman EL, Cohen HJ, Muss H, Rodin M, Panageas KS, Holland JC, Saltz L, Kris MG, Noy A, Gomez J, Jakubowski A, Hudis C, Kornblith AB. Developing a cancer-specific geriatric assessment: a feasibility study. Cancer. 2005 Nov 1;104(9):1998-2005. doi: 10.1002/cncr.21422. PMID 16206252
- [Background] Hurria A, Lichtman SM. Pharmacokinetics of chemotherapy in the older patient. Cancer Control. 2007 Jan;14(1):32-43. doi: 10.1177/107327480701400105. PMID 17242669
- [Background] Kimmick GG, Fleming R, Muss HB, Balducci L. Cancer chemotherapy in older adults. A tolerability perspective. Drugs Aging. 1997 Jan;10(1):34-49. doi: 10.2165/00002512-199710010-00004. PMID 9111706
- [Background] Talarico L, Chen G, Pazdur R. Enrollment of elderly patients in clinical trials for cancer drug registration: a 7-year experience by the US Food and Drug Administration. J Clin Oncol. 2004 Nov 15;22(22):4626-31. doi: 10.1200/JCO.2004.02.175. PMID 15542812
- [Background] Blackwell KL, Burstein HJ, Storniolo AM, Rugo H, Sledge G, Koehler M, Ellis C, Casey M, Vukelja S, Bischoff J, Baselga J, O'Shaughnessy J. Randomized study of Lapatinib alone or in combination with trastuzumab in women with ErbB2-positive, trastuzumab-refractory metastatic breast cancer. J Clin Oncol. 2010 Mar 1;28(7):1124-30. doi: 10.1200/JCO.2008.21.4437. Epub 2010 Feb 1. PMID 20124187

RESULTS

PARTICIPANT FLOW:
Groups:
- Age <=75; Age >75: Patients receive lapatinib ditosylate PO QD and trastuzumab IV once weekly OR once every 3 weeks. Courses repeat every 21 days in the absence of disease progression or unacceptable toxicity.
  Lapatinib: 250 mg tablets
  Trastuzumab: Intravenous injection
  laboratory biomarker analysis
  pharmacological study
Period: Overall Study
Arm/Group | Age <=75 | Age >75
Started | 30 | 10
Completed | 30 | 10
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Age ≤75: Participants 75 years of age and under receive lapatinib ditosylate 250mg PO QD and trastuzumab IV once weekly OR once every 3 weeks. Courses repeat every 21 days in the absence of disease progression or unacceptable toxicity.
- Age >75: Participants over 75 years of age receive lapatinib ditosylate 250mg PO QD and trastuzumab IV once weekly OR once every 3 weeks. Courses repeat every 21 days in the absence of disease progression or unacceptable toxicity.
- Total: Total of all reporting groups
Arm/Group | Age ≤75 | Age >75 | Total
Number analyzed (Participants) | 30 | 10 | 40
Age, Continuous [Mean (Full Range); unit: years] | 68 [60 to 75] | 84 [79 to 92] | 72 [60 to 92]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 30 | 9 | 39
  Male | 0 | 1 | 1
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 1 | 3
  Not Hispanic or Latino | 28 | 9 | 37
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 2 | 1 | 3
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 3 | 4
  White | 27 | 6 | 33
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 30 | 10 | 40
ECOG performance status [Count of Participants; unit: Participants]
  Fully active, able to carry on all pre-disease performance without restriction | 19 | 4 | 23
  Restricted in physically strenuous activity but ambulatory and able to do work of a light nature | 10 | 5 | 15
  Ambulatory and capable of selfcare but unable to do work activities; up and about >50% waking hours | 1 | 1 | 2

OUTCOME MEASURES:

1. Primary Outcome: Percent of Participants With Grade 3 or Higher Non-hematological Toxicities and Symptomatic Congestive Heart Failure
Description: Toxicities will be graded according to the National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) version 4.0. Rates and associated 95% exact Clopper and Pearson binomial confidence limits will be estimated for grade 3 or higher toxicities attributed to lapatinib or trastuzumab.
Time Frame: Until 30 days after last dose of treatment, an average of 8 months
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Age ≤75 | Age >75
Number analyzed (Participants) | 30 | 10
percentage of participants | 17 [6 to 35] | 30 [7 to 65]

2. Secondary Outcome: Percent of Participants With a Dose Modifications
Description: Rates and associated 95% exact Clopper and Pearson binomial confidence intervals will be estimated.
  A dose modification was defined as a hold (participant started the dose later than scheduled), reduction (subject was given a lower dose than originally scheduled), or discontinuation (subject stopped treatment) of lapatinib.
Time Frame: While on treatment, up to 4.5 years
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Age ≤75 | Age >75
Number analyzed (Participants) | 30 | 10
percentage of participants | 37 [20 to 56] | 60 [26 to 88]

3. Secondary Outcome: Number of Participants With Tumor Response Using Response Evaluation Criteria in Solid Tumors (RECIST)
Description: RECIST:
  Complete Response (CR): Disappearance of all target lesions. Lymph node CR is when the lymph node has decreased to less than 10mm in the short axis.
  Partial Response (PR): At least a 30% decrease in the sum of the longest diameter (LD) of target lesions, taking as reference the baseline sum LD.
  Progressive Disease (PD): At least a 20% increase in the sum of the LD of target lesions, taking as reference the smallest sum LD recorded since the treatment started (including the baseline scan if that is the smallest), and at least a 5mm increase or the appearance of new lesions.
  Stable Disease (SD): Neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for PD, taking as reference the smallest sum LD since the treatment started.
Time Frame: While on treatment, up to 4.5 years
Measure: Count of Participants; unit: Participants
Arm/Group | Age ≤75 | Age >75
Number analyzed (Participants) | 30 | 10
Participants
  Complete response (CR) | 0 | 1
  Partial response (PR) | 7 | 1
  Stable Disease (SD) | 6 | 3
  Progressive Disease | 12 | 0
  Not evaluable | 5 | 5

4. Secondary Outcome: Median Progression-free Survival (PFS)
Description: Median PFS and associated 95% exact Clopper and Pearson binomial confidence limits will be estimated across all ages per protocol plan.
  Progression is defined using RECIST v1.0, as at least a 20% increase in the sum of the LD of target lesions, taking as reference the smallest sum LD recorded since the treatment started (including the baseline scan if that is the smallest), and at least a 5mm increase or the appearance of new lesions.
Time Frame: From the date treatment begins until the first date on which recurrence, progression or death due to any cause, with an average follow up of 1 year.
Measure: Median (95% Confidence Interval); unit: months
Groups:
- Lapatinib and Trastuzumab: Participants receive lapatinib ditosylate 250mg PO QD and trastuzumab IV once weekly OR once every 3 weeks. Courses repeat every 21 days in the absence of disease progression or unacceptable toxicity.
Arm/Group | Lapatinib and Trastuzumab
Number analyzed (Participants) | 40
months | 2.7 [2.5 to 12]

5. Secondary Outcome: Median Overall Survival (OS)
Description: OS will be estimated using the product limit method of Kaplan and Meier across all ages per protocol plan.
Time Frame: Time from start of treatment to death due to any cause, with average follow up of 4.5 years
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Lapatinib and Trastuzumab
Number analyzed (Participants) | 40
months | 30.8 [17.9 to 39.9]

ADVERSE EVENTS:
Time Frame: On treatment plus 30 days following discontinuation of treatment, up to 4.5 years
Groups:
- Age > 75: Participants over 75 years of age receive lapatinib ditosylate 250mg PO QD and trastuzumab IV once weekly OR once every 3 weeks. Courses repeat every 21 days in the absence of disease progression or unacceptable toxicity.
Arm/Group | Age ≤75 | Age > 75
All-Cause Mortality (participants affected / at risk) | 19/30 | 7/10
Serious Adverse Events (participants affected / at risk) | 8/30 | 6/10
Other Adverse Events (participants affected / at risk) | 30/30 | 9/10
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Age ≤75 (N=30) | Age > 75 (N=10)
Diarrhea (Gastrointestinal disorders) | 3 | 1
Nausea (Gastrointestinal disorders) | 1 | 0
Vomiting (Gastrointestinal disorders) | 1 | 0
Bladder infection (Infections and infestations) | 0 | 1
Lung infection (Infections and infestations) | 0 | 1
Dehydration (Metabolism and nutrition disorders) | 1 | 1
Hyperglycemia (Metabolism and nutrition disorders) | 1 | 0
Hypoglycemia (Metabolism and nutrition disorders) | 1 | 0
Hypokalemia (Metabolism and nutrition disorders) | 0 | 1
Hyponatremia (Metabolism and nutrition disorders) | 0 | 1
Dizziness (Nervous system disorders) | 0 | 1
Edema cerebral (Nervous system disorders) | 1 | 0
Presyncope (Nervous system disorders) | 0 | 1
Seizure (Nervous system disorders) | 1 | 0
Vasovagal reaction (Nervous system disorders) | 1 | 0
Anxiety (Psychiatric disorders) | 1 | 0
Confusion (Psychiatric disorders) | 1 | 0
Psychosis (Psychiatric disorders) | 1 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Age ≤75 (N=30) | Age > 75 (N=10)
Anemia (Blood and lymphatic system disorders) | 12 | 3
Sinus bradycardia (Cardiac disorders) | 0 | 1
Vertigo (Ear and labyrinth disorders) | 0 | 2
Dry eye (Eye disorders) | 4 | 0
Watering eyes (Eye disorders) | 2 | 0
Abdominal distension (Gastrointestinal disorders) | 2 | 0
Abdominal pain (Gastrointestinal disorders) | 5 | 1
Bloating (Gastrointestinal disorders) | 4 | 0
Constipation (Gastrointestinal disorders) | 4 | 3
Diarrhea (Gastrointestinal disorders) | 27 | 8
Dry mouth (Gastrointestinal disorders) | 0 | 1
Dyspepsia (Gastrointestinal disorders) | 3 | 1
Flatulence (Gastrointestinal disorders) | 4 | 0
Gastroesophageal reflux disease (Gastrointestinal disorders) | 4 | 0
Mucositis oral (Gastrointestinal disorders) | 2 | 0
Nausea (Gastrointestinal disorders) | 11 | 5
Stomach pain (Gastrointestinal disorders) | 3 | 0
Vomiting (Gastrointestinal disorders) | 6 | 4
Edema limbs (General disorders) | 4 | 0
Fatigue (General disorders) | 18 | 6
Fever (General disorders) | 2 | 0
Flu like symptoms (General disorders) | 0 | 1
Localized edema (General disorders) | 3 | 1
Non-cardiac chest pain (General disorders) | 2 | 0
Pain (General disorders) | 13 | 2
Allergic reaction (Immune system disorders) | 2 | 0
Erythema (Infections and infestations) | 0 | 1
Lip infection (Infections and infestations) | 1 | 1
Lung infection (Infections and infestations) | 0 | 1
Nail infection (Infections and infestations) | 0 | 1
Papulopustular rash (Infections and infestations) | 2 | 1
Paronychia (Infections and infestations) | 5 | 3
Rash pustular (Infections and infestations) | 0 | 1
Skin infection (Infections and infestations) | 1 | 1
Upper respiratory infection (Infections and infestations) | 2 | 1
Urinary tract infection (Infections and infestations) | 2 | 1
Fall (Injury, poisoning and procedural complications) | 1 | 1
Alanine aminotransferase increased (Investigations) | 7 | 1
Alkaline phosphatase increased (Investigations) | 6 | 2
Aspartate aminotransferase increased (Investigations) | 6 | 3
Blood bilirubin increased (Investigations) | 4 | 2
Creatinine increased (Investigations) | 7 | 2
Ejection fraction decreased (Investigations) | 0 | 1
Lymphocyte count decreased (Investigations) | 3 | 1
Neutrophil count decreased (Investigations) | 0 | 1
Platelet count decreased (Investigations) | 3 | 0
Weight loss (Investigations) | 4 | 2
White blood cell decreased (Investigations) | 1 | 2
Anorexia (Metabolism and nutrition disorders) | 6 | 4
Hypercalcemia (Metabolism and nutrition disorders) | 3 | 0
Hyperglycemia (Metabolism and nutrition disorders) | 5 | 2
Hyperkalemia (Metabolism and nutrition disorders) | 2 | 0
Hypernatremia (Metabolism and nutrition disorders) | 3 | 0
Hypertriglyceridemia (Metabolism and nutrition disorders) | 2 | 0
Hypoalbuminemia (Metabolism and nutrition disorders) | 4 | 1
Hypocalcemia (Metabolism and nutrition disorders) | 3 | 0
Hypoglycemia (Metabolism and nutrition disorders) | 2 | 0
Hypokalemia (Metabolism and nutrition disorders) | 5 | 1
Hyponatremia (Metabolism and nutrition disorders) | 7 | 4
Arthralgia (Musculoskeletal and connective tissue disorders) | 4 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 8 | 0
Joint range of motion decreased (Musculoskeletal and connective tissue disorders) | 0 | 1
Leg cramping (Musculoskeletal and connective tissue disorders) | 0 | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 2 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 5 | 0
Dizziness (Nervous system disorders) | 4 | 0
Dysgeusia (Nervous system disorders) | 1 | 1
Headache (Nervous system disorders) | 6 | 2
Memory impairment (Nervous system disorders) | 0 | 1
Paresthesia (Nervous system disorders) | 2 | 0
Peripheral sensory neuropathy (Nervous system disorders) | 3 | 1
Presyncope (Nervous system disorders) | 1 | 1
Syncope (Nervous system disorders) | 0 | 1
Insomnia (Psychiatric disorders) | 2 | 0
Cystitis noninfective (Renal and urinary disorders) | 0 | 1
Allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 3 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 6 | 2
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 3 | 2
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 | 2
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 4 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Sleep apnea (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Sore throat (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Dry skin (Skin and subcutaneous tissue disorders) | 3 | 0
Nail ridging (Skin and subcutaneous tissue disorders) | 1 | 1
Pruritus (Skin and subcutaneous tissue disorders) | 4 | 1
Rash acneiform (Skin and subcutaneous tissue disorders) | 5 | 0
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 8 | 3
Hypertension (Vascular disorders) | 12 | 4
Thromboembolic event (Vascular disorders) | 2 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-04-19): https://cdn.clinicaltrials.gov/large-docs/10/NCT01273610/Prot_SAP_000.pdf